CLINICAL TRIAL: NCT05430048
Title: Preoperative Nasal Desmopressin Versus Oral Bisoprolol for Controlling Bleeding and Improving Surgical Field During Unilateral Functional Endoscopic Sinus Surgery
Brief Title: Nasal Desmopressin Versus Oral Bisoprolol for Controlling Bleeding During Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba M Fathi, Dr. Heba M Fathi, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9262
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-06

CONDITIONS: Bleeding
Keywords: Desmopressin ,bisoprolol,Sinus Surgery
MeSH Terms: conditions — Hemorrhage | interventions — Bisoprolol

STUDY DESIGN:
Intervention Model Description: comparing Preoperative Nasal Desmopressin versus Oral Bisoprolol for Controlling Bleeding and Improving Surgical Field during Unilateral Functional Endoscopic Sinus Surgery
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desmopressin group (Group D) (Active Comparator): patients will received single puff (10 μg) of nasal desmopressin in the nasal cavity at the side of surgery 30 min preoperative.
  Interventions: Drug: nasal Desmopressin
- Bisoprolol group (group B) (Active Comparator): patients will receive Oral bisoprolol 2.5 mg (Concor 2.5 mg; Merck/Amoun) 90 min preoperative.
  Interventions: Drug: nasal Desmopressin

INTERVENTIONS:
Drug: nasal Desmopressin — compare the effect of nasal desmopressin versus oral bisoprolol for controlling bleeding and improving surgical field clarity during functional endoscopic sinus surgery.
  Other Names: oral Bisoprolol

SUMMARY:
Functional endoscopic sinus surgery (FESS) is well established for treatment of chronic rhinosinusitis and nasal polyps. Masking of the surgical field can lead to severe complication as tissue injury, increase post-operative adhesions and scarring and even severe orbital and brain injury In the current study we will investigate the effect of nasal desmopressin versus oral bisoprolol for controlling bleeding and improving surgical field clarity during functional endoscopic sinus surgery

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is well established for treatment of chronic rhinosinusitis and nasal polyps.

The nasal mucosa at the site of surgery is very sensitive to sympathetic stimulation which Cause intraoperative hypertension and tachycardia. It is also highly vascular and can bleed easily, so Compromise the visual clarity of the surgical field. Masking of the surgical field can lead to severe complication as tissue injury, increase post-operative adhesions and scarring and even severe orbital and brain injury. Multiple techniques have been discussed to improve the surgical field in endoscopic sinus surgery, including the use of bipolar diathermy, topical vasoconstrictors, and induced hypotension, However none of them has provided optimal surgical condition.

Desmopressin (1 deamino 8 D argininevasopressin) is a synthetic analog of the antidiuretic hormone L arginine vasopressin. It was used in mild to moderate hemophilia, von Willebrand's disease, and other acquired platelet deficiencies to increases plasma concentrations of tissue plasminogen activator and endothelial factor VIII. Intravenous use was proved to decrease intraoperative bleeding during spine surgery, facial plastic surgeries, septo-rhinoplasty and FESS. Intranasal spray used effectively to reduce bleeding and improves the surgical field during FESS.

The short acting β-adrenergic receptor antagonist such as labetalol, metoprolol and esmolol have been successfully used for lowering blood pressure, decreasing bleeding and improving surgical field.

Bisoprolol, has the advantage of longer acting. Bisoprolol has a higher degree of β1-selectivity compared to other β1-selective beta blockers such as atenolol, metoprolol, and betaxolol. It was approved for medical use in the United States in 1992. Bisoprolol inhibits renin secretion by about 65% and tachycardia by about 30%.

In the current study we will investigate the effect of nasal desmopressin versus oral bisoprolol for controlling bleeding and improving surgical field clarity during functional endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria: patients scheduled for unilateral functional endoscopic sinus surgery, aged between 21 - 60 years, both genders, ASA grade I - II and body mass index 25-30 kg/m -

Exclusion Criteria: Patients with acute decompensated heart failure, Peripheral vascular disease, hypertension, heart block, Asthma, bleeding disorders, coronary disease, compromised renal or hepatic function, hyponatremia , pregnancy or history of allergy to the study drugs and those on anti-platelet, anticoagulant or B blocker drugs.

-

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
the volume of blood loss in cubic centimeter | during surgeries
  the volume of blood loss in cubic centimeter calculating as (the volume of fluid in the suction bottle after deduction of normal saline volume that will be used for endoscopic scrub, plus the volume of soaked cotton strip (fully soaked will be estimated to contain 5 ml of blood and a partially soaked will be estimated to contain 2.5 ml)

SECONDARY OUTCOMES:
The quality of surgical field | measured every 15 minutes from beginning of surgery until the end of surgery
  The quality of surgical field using Boezaart surgical field grading scale

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Fathi, Principal Investigator — Zagazig University
Locations (1):
- Heba M Fathi, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No